CLINICAL TRIAL: NCT06443307
Title: A Prospective, Multi-cohort, National Multicenter Real-world Study to Evaluate the Efficacy and Safety of Liposome Irinotecan
Brief Title: Real-world Study to Evaluate the Efficacy and Safety of Liposome Irinotecan
Status: Recruiting | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Other Study IDs: CSPC-DEY-CRC-K02
Record Dates: First submitted 2024-05-15; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Cancer; Solid Tumor
MeSH Terms: conditions — Colorectal Neoplasms | interventions — irinotecan sucrosofate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Second-line treatment for colorectal cancer: Cohort 1 is a concurrent control design, including patients treated with irinotecan liposome (Nal-IRI) or irinotecan (IRI) plus fluorouracils as second-line treatment for metastatic colorectal cancer.
  Interventions: Drug: Irinotecan Liposome
- Posterior line treatment of colorectal cancer: Cohort 2 is a Simon two-stage design, is planned to include patients who are treated with a NAL-IRI based combination regimen and have used IRI as a late-line treatment for metastatic colorectal cancer.
  Interventions: Drug: Irinotecan Liposome
- Neoadjuvant therapy for colorectal cancer: Cohort 3 is a single-arm design and planned to enroll patients who received Nal-IRI+ oxaliplatin + fluorouracils as neoadjuvant chemotherapy for colorectal cancer.
  Interventions: Drug: Irinotecan Liposome
- Patients with non-pancreatic and non-colorectal cancer received second-line or above treatment: Cohort 4 is a single-arm design and is planned to enroll patients who are treated with the NAL-IRI containing regimen as second-line or beyond treatment for nonpancreatic, noncolorectal cancers.
  Interventions: Drug: Irinotecan Liposome

INTERVENTIONS:
Drug: Irinotecan Liposome — The experimental group will collect data from patients treated with Nal-IRI as the chemotherapy regimen. It is recommended to use according to the label, clinical practice shall prevail.

SUMMARY:
This study is a prospective, multicenter, real-world study. There are four cohorts. Cohorts 1-3 include second-line, posterior-line, and neoadjuvant colorectal cancer patients, respectively. Cohort 4 include patients with the exception of those with pancreatic and colorectal cancer. As this study is a real-world investigation, treatment procedures, visit schedules, and examinations will be based on the routine clinical practice of physicians. Through the above cohort, the efficacy and safety of irinotecan liposome are comprehensively observed.

ELIGIBILITY:
Inclusion Criteria:

1. Cohort 1:

   * Patients with histologically or cytopathologically confirmed colorectal adenocarcinoma who were diagnosed with unresectable metastatic disease.
   * Known to be pMMR/MSS or MMR/MS status unknown.
   * Prior first-line systemic oxaliplatin - and fluorouracils-based therapy for metastatic disease progressed.
   * Patients had not received IRI or Nal-IRI during the treatment phase of metastatic disease.
   * Patients were scheduled to receive Nal-IRI plus fluorouracils or IRI plus fluorouracils chemotherapy regimens as second-line systemic therapy.
2. Cohort 2:

   * Patients with histologically or cytopathologically confirmed colorectal adenocarcinoma who were diagnosed with unresectable metastatic disease;
   * Known to be pMMR/MSS or MMR/MS status unknown.
   * Patients had received ≤ 3 lines of previous treatment for metastatic disease.
   * Progression of metastatic disease after treatment with an IRI-containing regimen (no limit on the number of IRI treatment lines).
   * The patient had not previously received Nal-IRI and was scheduled to receive a systemic Nal-IRI containing chemotherapy regimen as palliative treatment.
   * Have at least one measurable lesion according to RECIST v1.1.
3. Cohort 3:

   * High-risk (CRS score 3-5) synchronous liver metastatic colorectal adenocarcinoma with ≤5 liver metastases, confirmed by histopathology or cytopathology, and planned resection.
   * Known to be pMMR/MSS or MMR/MS status unknown.
   * The patient was scheduled to receive Nal-IRI+ oxaliplatin + fluorouracils chemotherapy regimen as neoadjuvant therapy.
4. Cohort 4:

   * Non pancreatic cancer and non colorectal cancer patients confirmed by histopathology and/or cytology.
   * Have received at least one systemic treatment for unresectable diseases;
   * Plan to receive a systemic treatment regimen containing Nal IRI;
   * At least one measurable lesion (according to RECIST v1.1);

Exclusion Criteria:

Cohort 1-4:

* Treatment with an immune checkpoint inhibitor (e.g., pembrolizumab, nivolumab) was planned during chemotherapy.
* Allergy to irinotecan or liposomal irinotecan and its excipients is known.
* Female patients known to be pregnant or lactating.
* Other patients who were deemed by the investigator to be ineligible for enrollment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study was a prospective, multicenter real-world study with four cohorts. Cohort 1 include patients as second-line treatment for metastatic colorectal cancer. Cohort 2 include patients as a late-line treatment for metastatic colorectal cancer. Cohort 3 include patients as neoadjuvant chemotherapy for colorectal cancer.
  Cohort 4 include patients as second-line or beyond treatment for nonpancreatic, noncolorectal cancers. Through the above cohort, the efficacy and safety of irinotecan liposome are comprehensively observed.
Sampling Method: Non-Probability Sample
Enrollment: 933 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade ≥3 adverse events assessed by CTCAE 5.0 (Cohort 1) | Assessed except to 10 months.
  To investigate the safety with Nal-IRI and IRI.
Objective response rate (Cohort 2 and 4) | From initial medication to the date of first documented progression or end of medication. Assessed up to 6 months.
  To investigate antitumor efficacy of Nal-IRI, proportion of patients with complete (CR) or partial response (PR) assessed by RECIST v1.1.
R0 resection rate (Cohort 3) | From initial medication to the date of first documented progression or end of medication. Assessed up to 6 months.
  To assess surgical conversion rates in patients who could be surgically resected.

SECONDARY OUTCOMES:
Objective response rate (Cohort 1) | From initial medication to the date of first documented progression or end of medication. Assessed up to 6 months.
  To investigate antitumor efficacy of Nal-IRI, proportion of patients with complete (CR) or partial response (PR) assessed by RECIST v1.1.
Disease control rate (Cohort 1,2,4) | From initial medication to the date of first documented progression or end of medication.Assessed up to 6 months.
  To investigate antitumor efficacy of Nal-IRI, proportion of patients with complete , partial or stable response (SD) assessed by RECIST v1.1.
Progression free survival (Cohort 1,2,4) | From initial medication to the date of first documented progression or date of death from any cause, whichever came first. Assessed up to 24 months.
  To investigate antitumor efficacy of study. From initial medication to the date of first documented progression or end of medication, whichever came first.
Overall survival (Cohort 1,2,4) | From initial medication to the date of death from any cause. Assessed up to 42 months.
  To investigate antitumor efficacy of Nal-IRI. From initial medication to the date of death from any cause.
Incidence of adverse events and severity of adverse events as assessed by CTCAE 5.0 (Cohort 1,2,3,4) | Assessed except to 24 months.
  To assess the incidence and severity of adverse events in combination regimens.
Pathological complete response rate (Cohort 3) | After treatment and surgery, assessed up to 6 months.
  To investigate the effect of Nal-IRI.
Event-free survival (Cohort 3) | The time from enrollment to any event, including death, disease progression, or switch to a treatment, occurred first. Assessed up to 12 months.
  To investigate the effect of Nal-IRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China